CLINICAL TRIAL: NCT03459690
Title: EEG Changes With Meditation: A Proposal to Analyze EEG Changes With a Simple, Online, Guided Meditative Tool.
Brief Title: EEG Changes With Guided Online Meditation
Acronym: IKEEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Director, Center for Anesthesia Research Excellence, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018P000040
Record Dates: First submitted 2018-02-14; First posted 2018-03-09 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-09

CONDITIONS: Meditation
Keywords: Meditation, EEG
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Intervention Model Description: This is a prospective trial enrolling healthy volunteers, including novice meditators and experienced meditators. Subjects will undergo an EEG at baseline and again after 6 weeks. During the 6 weeks, subjects will be asked to meditate twice a day, 12 minutes each time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experienced meditators (Experimental): Meditation ≥ 30 min per day for at least 5 days per week over the past 1 year
  Interventions: Behavioral: Meditation; Device: Enobio 32- EEG machine
- Novice meditators (Experimental): No meditation practice in the previous year and < 20 entire lifetime hours
  Interventions: Behavioral: Meditation; Device: Enobio 32- EEG machine

INTERVENTIONS:
Behavioral: Meditation — Isha Kriya meditation is simple meditation practice which can be easily learned by employing online guided tools. Isha Kriya meditation requires approximately 12 minutes, twice a day of practice. This regimen was chosen because of its simplicity making it an excellent way to introduce meditation to beginners. Isha Kriya does not incorporate a spiritual or religious focus.
Device: Enobio 32- EEG machine — This study utilizes the Enobio 32 EEG device made by Neuroelectrics (an FDA-cleared 24-bit EEG data reader which is a wearable wireless device) to analyze EEG changes after subjects have undergone meditation. This study does not evaluate the Enobio device, and the IRB of record approved an Investigational Device Exemption for this study.

SUMMARY:
Simple meditation and EEG changes

DETAILED DESCRIPTION:
This is a prospective trial enrolling healthy volunteers, including novice meditators and experienced meditators. Subjects will undergo an EEG at baseline and again after 6 weeks. During the 6 weeks, subjects will be asked to meditate twice a day, at least 12 minutes each time.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Novice or expert meditator

Novice meditator: No meditation practice in the previous year and < 20 entire lifetime hours

Expert meditator: Meditation ≥ 30 min per day for at least 5 days per week over the past 1 year

Exclusion Criteria:

1. History of any neurological condition (i.e. Parkinson's disease, Alzheimer's disease, Huntington's disease, brain tumors, brain surgery, or multiple sclerosis)
2. History of depression, currently being treated with antidepressants
3. History of any psychiatric disorder, within last 5 years (i.e. anxiety, psychosis, posttraumatic stress disorder, attention deficit hyperactive disorder)
4. Current use of cognition-enhancing medications
5. Active history (within the last 5 years) of alcohol or drug abuse (> 10 drinks per week)
6. History (within the last 5 years) of stroke/aneurysm
7. Recent history (< 3 months) of seizures
8. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Experienced Meditators: Meditation ≥ 30 min per day for at least 5 days per week over the past 1 year
  Meditation: . IK is a meditation that can be learned quickly and requires approximately 12 minutes, twice a day of practice. This regimen was chosen because of its simplicity making it an excellent way to introduce meditation to beginners. IK does not incorporate a spiritual or religious focus
- Novice Meditators: No meditation practice in the previous year and < 20 entire lifetime hours
  Meditation: . IK is a meditation that can be learned quickly and requires approximately 12 minutes, twice a day of practice. This regimen was chosen because of its simplicity making it an excellent way to introduce meditation to beginners. IK does not incorporate a spiritual or religious focus
Period: Overall Study
Arm/Group | Experienced Meditators | Novice Meditators
Started | 4 | 9
Completed | 3 | 7
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Of the 13 participants enrolled in the study 2 participants requested withdrawal and 1 was lost to follow up, resulting in 7 novice meditators and 3 experienced meditators who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experienced Meditators | Novice Meditators | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (9.04) | 34.75 (18.84) | 47.58 (15.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 7 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 4 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With EEGs to Measure Changes in Wave Oscillations
Description: Number of participants who had EEGs to measure qualitative changes in wave oscillations
Time Frame: 6 weeks
Population: Of the 13 participants enrolled in the study 2 participants requested withdrawal and 1 was lost to follow up, resulting in 7 novice meditators and 3 experienced meditators who completed the study. Following data cleaning for signal strength & intensity among these 10 participants, only 7 participants (3 Experienced & 4 Novice) had usable data for analysis.
Measure: Number; unit: Participants with Evaluable EEGs
Arm/Group | Experienced Meditators | Novice Meditators
Number analyzed (Participants) | 3 | 7
Participants with Evaluable EEGs | 3 | 4

2. Secondary Outcome: Number of Participants With Evaluable EEGs to Measure Changes in Wave Amplitude
Description: Number of participants who had evaluable EEGs to measure qualitative changes in wave amplitude
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experienced Meditators | Novice Meditators
Number analyzed (Participants) | 3 | 7
Participants | 3 | 4

3. Secondary Outcome: Number of Participants With Evaluable EEGs to Measure Changes in Wave Latency
Description: Number of participants who had evaluable EEGs to measure qualitative changes in wave latency
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experienced Meditators | Novice Meditators
Number analyzed (Participants) | 3 | 7
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Experienced Meditators | Novice Meditators
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 0/4 | 0/9

LIMITATIONS AND CAVEATS:
1. The total number of participants enrolled in the study (n=13) was small, which means that the strength of the statistical test will be low.
2. Participant numbers with evaluable EEG was even smaller. Hence, group level analysis could not be performed in the study and the effects were assessed at an individual level.
3. Technical issues such as bad channels, corrupt data files and missing files marred the collected data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03459690/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03459690/ICF_001.pdf